CLINICAL TRIAL: NCT01424982
Title: Phase II Study of Combination of Hyper-CVAD and Ponatinib in Patients With Philadelphia (PH) Chromosome Positive and/or BCR-ABL Positive Acute Lymphoblastic Leukemia (ALL)
Brief Title: Combination Chemotherapy and Ponatinib Hydrochloride in Treating Patients With Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0030; NCI-2011-02941 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0030 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2011-08-24; First posted 2011-08-29 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Lymphoblastic Leukemia; Adult Acute Lymphoblastic Leukemia in Complete Remission; B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Philadelphia Chromosome Positive; Untreated Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Methotrexate; merphos; ponatinib; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (combination chemotherapy, ponatinib hydrochloride) (Experimental): See Detailed Description.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Drug: Ponatinib; Drug: Ponatinib Hydrochloride; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Ponatinib — Given PO
  Other Names: AP-24534; AP24534
Drug: Ponatinib Hydrochloride — Given PO
  Other Names: AP24534 HCl; Iclusig
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Vincristine — Given IV
  Other Names: LEUROCRISTINE; VCR; Vincrystine
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies the side effects and how well combination chemotherapy and ponatinib hydrochloride work in treating patients with acute lymphoblastic leukemia. Drugs used in chemotherapy, such as cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ponatinib hydrochloride may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy and ponatinib hydrochloride may be an effective treatment for acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the clinical efficacy (event-free survival) of an intensive short-term chemotherapy regimen (hyperfractionated cyclophosphamide-vincristine sulfate-Adriamycin [doxorubicin hydrochloride]-dexamethasone [hyper-CVAD] program) given in combination with the tyrosine kinase inhibitor ponatinib hydrochloride (ponatinib) for Philadelphia (Ph)-positive and/or BCR-ABL-positive acute lymphoblastic leukemia (ALL).

II. To evaluate other clinical efficacy endpoints (overall response rate and survival) and safety of the regimen.

OUTLINE:

ODD CYCLES (1, 3, 5, and 7): Patients receive cyclophosphamide intravenously (IV) over 3 hours every 12 hours on days 1-3, doxorubicin hydrochloride IV continuously over 24 hours on day 4, vincristine sulfate IV over 30 minutes on days 1 and 11, dexamethasone IV over 30 minutes or orally (PO) once daily (QD) on days 1-4 and 11-14, and ponatinib hydrochloride PO QD on days 1-14 of cycle 1 and continuously in cycles 3, 5, and 7. Patients with CD20 expression may also receive rituximab IV on days 1 and 11 of cycle 1 and 3. Treatment repeats every 3-4 weeks for up to 8 cycle in the absence of disease progression or unacceptable toxicity.

EVEN CYCLES (2, 4, 6, and 8): Patients receive methotrexate IV over 24 hours on day 1, ponatinib hydrochloride PO QD continuously, and cytarabine IV over 3 hours every 12 hours on days 2 and 3. Patients with CD20 expression may also receive rituximab IV on days 1 and 8 of cycle 2 and 4. Treatment repeats every 3-4 weeks for up to 8 cycle in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive vincristine sulfate IV on day 1, prednisone PO daily on days 1-5, and ponatinib hydrochloride PO QD on days 1-28. Cycle repeat every 28 days for 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following:

  * Previously untreated Ph-positive ALL [either t(9;22) and/or bcr-abl positive] (includes patients initiated on first course of hyper-CVAD before cytogenetics known) or with lymphoid accelerated or blast phase chronic myelogenous leukemia (CML)
  * Previously treated Ph-positive ALL or CML (in accelerated phase or blast phase), after 1-2 courses of chemotherapy with or without other tyrosine kinase inhibitors (TKIs)

    * If they achieved complete response (CR), they are assessable only for event-free and overall survival, or
    * If they failed to achieve CR, they are assessable for CR, event-free, and overall survival
* Performance status ≤ 2 (Eastern Cooperative Oncology Group [ECOG] scale, Appendix E)
* Adequate liver function as defined by the following criteria:
* Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome
* Alanine aminotransferase (ALT) ≤ 2 x ULN
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Adequate pancreatic function as defined by the following criteria:
* Serum lipase and amylase ≤ 1.5 x ULN
* For females of childbearing potential, a negative pregnancy test must be documented prior to randomization
* Female and male patients who are fertile must agree to use an effective form of contraception with their sexual partners from randomization through 4 months after the end of treatment
* Adequate cardiac function as assessed clinically by history and physical examination
* Signed informed consent

Exclusion Criteria:

* Active serious infection not controlled by oral or intravenous antibiotics
* History of acute pancreatitis within 1 year of study or history of chronic pancreatitis
* History of alcohol abuse
* Uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL)
* Active secondary malignancy other than skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year
* Active grade III-V cardiac failure as defined by the New York Heart Association criteria
* Clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

  * Any history of myocardial infarction (MI), stroke, or revascularization
  * Unstable angina or transient ischemic attack prior to enrollment
  * Congestive heart failure prior to enrollment, or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards prior to enrollment
  * Diagnosed or suspected congenital long QT syndrome
  * Any history of clinically significant atrial or ventricular arrhythmias (such as atrial fibrillation, ventricular tachycardia, ventricular fibrillation, or torsades de pointes) as determined by the treating physician
  * Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 470 msec) unless corrected after electrolyte replacement
  * Any history of venous thromboembolism including deep venous thrombosis or pulmonary embolism
  * Uncontrolled hypertension (diastolic blood pressure > 90 mmHg; systolic > 140 mmHg); patients with hypertension should be under treatment on study entry to effect blood pressure control
* Patients currently taking drugs that are generally accepted to have a risk of causing torsades de pointes (unless these can be changed to acceptable alternatives)
* Taking any medications or herbal supplements that are known to be strong inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) within at least 14 days before the first dose of ponatinib
* Prior history of treatment with ponatinibfor > 1 month; patient who has been treated with ponatinib for 1 month prior starting the treatment is eligible
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator; patient who has been treated with ponatinib for 1 month prior starting the treatment is eligible
* Pregnant and lactating women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception; women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months; in addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* Patients with documented significant pleural or pericardial effusions unless they are thought to be secondary to their leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2011-10-05 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | The time from the start of the treatment until any failure (resistant disease, relapse, or death), assessed up to 24 months
  Kaplan-Meier survival curves will be constructed.

SECONDARY OUTCOMES:
Complete response rate | Up to 24 months after completion of study treatment
  Complete response is defined as achieving bone marrow blasts =< 5% AND platelets >= 100 AND absolute neutrophil count >= 1000 within 3 courses of treatment. The method of Thall, Simon, and Estey will be employed to perform short-term interim efficacy. Response rate and its corresponding 95% confidence interval will be provided at the end of the study.
Incidence of grade 3-4 toxicity according to the M.D. Anderson Leukemia-specific Adverse Event Recording and Reporting Guidelines | Up to 24 months
  The method of Thall, Simon, and Estey will be employed to perform short-term interim safety monitoring. Will be summarized in frequency tables or in the form of mean, standard deviation, and range where appropriate. Toxicity rate and its corresponding 95% confidence interval will be provided at the end of the study.
Overall survival | Up to 24 months after completion of study treatment
  Kaplan-Meier survival curves will be constructed. Survival rates at specific time points will be estimated along with corresponding 95% confidence intervals.
Disease-specific survival | Up to 24 months after completion of study treatment
  Kaplan-Meier survival curves will be constructed. Survival rates at specific time points will be estimated along with corresponding 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kantarjian H, Short NJ, Jain N, Sasaki K, Huang X, Haddad FG, Khouri I, DiNardo CD, Pemmaraju N, Wierda W, Garcia-Manero G, Kebriaei P, Garris R, Loghavi S, Jorgensen J, Kwari M, O'Brien S, Ravandi F, Jabbour E. Frontline combination of ponatinib and hyper-CVAD in Philadelphia chromosome-positive acute lymphoblastic leukemia: 80-months follow-up results. Am J Hematol. 2023 Mar;98(3):493-501. doi: 10.1002/ajh.26816. Epub 2023 Jan 4. PMID 36600670
- [Derived] Jabbour E, Short NJ, Ravandi F, Huang X, Daver N, DiNardo CD, Konopleva M, Pemmaraju N, Wierda W, Garcia-Manero G, Sasaki K, Cortes J, Garris R, Khoury JD, Jorgensen J, Jain N, Alvarez J, O'Brien S, Kantarjian H. Combination of hyper-CVAD with ponatinib as first-line therapy for patients with Philadelphia chromosome-positive acute lymphoblastic leukaemia: long-term follow-up of a single-centre, phase 2 study. Lancet Haematol. 2018 Dec;5(12):e618-e627. doi: 10.1016/S2352-3026(18)30176-5. PMID 30501869
- [Derived] Jabbour E, Kantarjian H, Ravandi F, Thomas D, Huang X, Faderl S, Pemmaraju N, Daver N, Garcia-Manero G, Sasaki K, Cortes J, Garris R, Yin CC, Khoury JD, Jorgensen J, Estrov Z, Bohannan Z, Konopleva M, Kadia T, Jain N, DiNardo C, Wierda W, Jeanis V, O'Brien S. Combination of hyper-CVAD with ponatinib as first-line therapy for patients with Philadelphia chromosome-positive acute lymphoblastic leukaemia: a single-centre, phase 2 study. Lancet Oncol. 2015 Nov;16(15):1547-1555. doi: 10.1016/S1470-2045(15)00207-7. Epub 2015 Sep 30. PMID 26432046
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org